CLINICAL TRIAL: NCT04069364
Title: Systematische Untersuchung Zum Einfluss Von Selbsthilfe Auf Die Subjektive Belastung Bei Chronischem Tinnitus
Brief Title: Systematic Assessment of Self-help Tools for the Management of Chronic Tinnitus
Acronym: TinnitusTips
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Winfried Schlee, Head of eHealth Group, University Hospital Regensburg
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-544-101
Record Dates: First submitted 2019-04-29; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: TinnitusTipps — Self-helf tips for managing chronic tinnitus will be given via smartphones.

SUMMARY:
With this study we want to investigate the impact of self-help tools on the subjective tinnitus distress in chronic tinnitus patients.

Furthermore, we want to investigate the influence of personal characteristics on the individual tinnitus improvement.

DETAILED DESCRIPTION:
A smart-phone app running on iOS devices will be used to give self-help tips to the chronic tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic tinnitus, duration at least 6 monhts

Exclusion Criteria:

* acute psychosis, depression, substance abuse
* psychopharmaca
* epilepsy or other disease of the central nervous system
* other tinnitus treatments in the last 3 months
* drug, medication or alcohol abuse in the last 12 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of Tinnitus Handicap Inventory | Before, after 4 months, and after 6 months
  Questionnaire
Change of Tinnitus Numeric Rating Scale | Before, after 4 months, and after 6 months
  Questionnaire
Change Clinical Global Impression | Before, after 4 months, and after 6 months
  Questionnaire

SECONDARY OUTCOMES:
Change of WHO Quality of Life | Before, after 4 months, and after 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided